CLINICAL TRIAL: NCT01279551
Title: Topical Application of GTN 0.4% in the Treatment of Anismus Following Stapled Haemorrhoidopexy
Acronym: TAGASH
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DS-003
Record Dates: First submitted 2011-01-18; First posted 2011-01-19 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2011-01

CONDITIONS: Pain After Stapled Haemorrhoidopexy
MeSH Terms: interventions — Ointments

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- GTN (Experimental): In this arm the investigators administer local application of 0.4% nitroglycerin ointment and ketorolac tromethamine 10 mg
  Interventions: Drug: 0.4% nitroglycerin ointment
- Control (Active Comparator): In this arm the investigators administer local application of lidocaine cloridrato 2.5% and ketorolac tromethamine 10 mg.
  Interventions: Drug: lidocaine cloridrato 2.5% ointment

INTERVENTIONS:
Drug: 0.4% nitroglycerin ointment — Local endoanal application 2 times a day
  Other Names: Rectogesic
  Arms: GTN
Drug: lidocaine cloridrato 2.5% ointment — Local endoanal application of lidocaine cloridrato 2.5% ointment 2 times a day
  Other Names: Luan
  Arms: Control

SUMMARY:
This study wants demonstrate that the use of 0.4% nitroglycerin ointment can reduce the postoperative pain related to anorectal spasm (anismus) while performing a stapled haemorrhoidopexy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic II-III grade haemorrhoids and rectal mucosal prolapse
* Adults aged ≤ 75, male or female

Exclusion Criteria:

* Concomitant ano-rectal disease (fissure, fistula, abscess, inflammatory bowel disease, rectal cancer)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2004-01; Primary Completion 2010-09 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Postoperative pain related to upper anal canal pressure increasing (yes or no) | from the intervention to 1 month
  To evaluate if the pain post stapled haemorrhoidopexy is related to an increased anal resting pressure or not. The presence of anorectal spasm was assessed by clinical examination and anorectal manometry
Postoperative pain remission | from 1 to 90 days after intervention
  To assess postoperative pain remission
Postoperative anal resting pressure at pain remission | from 1 to 90 days after intervention
  We evaluate with anorectal manometry the anal resting pressure at the time of pain remission

SECONDARY OUTCOMES:
Duration of therapy | from 1 to 90 days after intervention
  To evaluate how many days of therapy are needed to obtain pain remission
Use of additional analgesic | from 1 to 90 days to intervention
  To evaluate the use of additional drugs respect to standard therapy
Postoperative pain intensity | from 1 to 90 days after intervention
  To evaluate the intensity of postoperative pain assessed by VAS (visual analogue scale)
Patients satisfaction | 45 days after intervention
  To evaluate the satisfaction of the patients, assessed by a questionnaire (scale from 1 to 5)

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Saverio Mari, MD, Principal Investigator — Oneday-Day Surgery Unit, II Faculty of Medicne and Surgery, Sapienza University of Rome; Luigi Masoni, MD, Study Chair — Oneday-Day Surgery Unit, II Faculty of Medicne and Surgery, Sapienza University of Rome
Locations (1):
- Oneday-Day Surgery Unit, II Faculty of Medicne and Surgery, Sapienza University of Rome, Rome, Italy

REFERENCES:
- [Derived] Mari FS, Nigri G, Dall'Oglio A, Cosenza UM, Milillo A, Terrenato I, Pancaldi A, Brescia A. Topical glyceryl trinitrate ointment for pain related to anal hypertonia after stapled hemorrhoidopexy: a randomized controlled trial. Dis Colon Rectum. 2013 Jun;56(6):768-73. doi: 10.1097/DCR.0b013e31828b282c. PMID 23652752